# Journey of Transformation Curriculum for Native American Adolescents (JOT)

## NCT05274217

Teresa Evans-Campbell, PhD

**Assent Form** 

IRB Approved 09-07-2022

#### UNIVERSITY OF WASHINGTON

# ASSENT TO RESEARCH JOURNEY OF TRANSFORMATION

### Researchers:

 Tessa Evans-Campbell, Associate Professor, School of Social Work, University of Washington, 206-849-9463, tecamp@uw.edu

#### Researcher's statement:

My name is [identify yourself to the child by name].

We are asking you to be in a research study because we are trying to learn more about a new curriculum that will be available to freshmen. The lessons will include traditional storytelling and other Native American cultural arts activities (i.e., drum making, film making, field trips), as well as Traditional Ecological Knowledge (TEK) activities. We would like to know how well the curriculum explains leadership skills, Native American cultural arts, the natural environment, and promotes healthy decision-making around health and relationships.

If you agree to be in this study, your health class will be assigned by chance [randomly, like flipping a coin] to start the research curriculum in the fall or to start the research program in the winter. During the semester you participate in the program, the class will:

<u>Week 1</u>. Take a 30-40 minute online survey about healthy relationships, drug use, youth leadership skills and connecting with Native communities.

<u>Weeks 1-3</u>. Meet to set goals around health, healthy relationships and how to reduce or avoid alcohol, tobacco, or other drug use.

Weeks 1-8 (months 1-2). As part of your class, attend about 16 health sessions on healthy behaviors and health promotion. Learn new skills around youth leadership, storytelling, and traditional health practices. The sessions will highlight connecting to tribal traditions.

Month 3. Take an online check-in survey via a link sent to your email address.

Month 6. Take an online check-in survey via a link sent to your email address.

Month 12. Take an online check-in survey via a link sent to your email address.

#### **Optional after school activities**

<u>Week 9- 16 (months 3-4)</u>. Attend a once-a-month activity to help build leadership skills. Activities are between 1-2 hours after school and include drum making, film making, creating a storytelling vest that incorporates your own cultural symbols, and up to two outdoor field trips. The field trips are to places of cultural significance near the school and involve a 30-45 minute hike.

<u>Week 16 (month 4)</u>. Meet with a mentor to revise your goals for health and community leadership.

<u>Week 9 -24 (months 3 - 6)</u>. Attend a 2-hour digital storytelling training and three-monthly planning sessions to prepare for an optional digital storytelling leadership night. Your story can be about what you have learned about health promotion, traditional health practices, and to celebrate your health leadership journey.

<u>Week 25 (month 6)</u>. Attend the leadership night and present your digital stories if you would like. Help prepare a traditional feast and giveaway that will honor your community culture and values.

<u>Health survey questions</u>. The survey will ask questions about your health behaviors, connection to others, and cultural connections as well as substance use and sexual health. Examples of some of the most sensitive questions you will be asked to answer in the survey are: "During last 12 months have you had sexual intercourse with other youth" and "During the past month, what was the most you had to drink in any one day." Your answers will be directly linked to a study ID number and not directly linked to your name. The study team will not share your survey responses with your parents. <u>You are</u> free to not answer any questions that you do not want to answer.

**Your participation in this study is voluntary.** Participation throughout this research study is completely voluntary and confidential. You are free to withdraw from this study at any time without any consequences.

<u>Potential risks</u>: Some of the questions will ask about thoughts, feelings, and personal difficulties that may be private and feel sensitive. You may feel embarrassed or anxious if you choose to disclose personal information. You will be asked about substance use, trauma exposure, and your health behaviors and about potentially illegal behaviors such as substance use. These questions may make you feel uncomfortable, bring back stressful or upsetting memories or seem intrusive. If you experience an increase in emotional distress related to your participation in the project, please let study staff know so that we can provide appropriate support.

You may also worry about people finding out what you say in the survey or during the study activities. There is a small risk of someone outside the study finding out personal information, but we have taken steps to reduce this risk. We will keep all data (your answers to the surveys) confidential and will only share this outside of the study team when it is necessary. For example, your answers are encrypted and they are not connected to your name. Instead, we use a unique code to link your name and the data. The link file is on a secure server and is password protected.

During the optional outdoor activities, you may feel environmentally-based discomfort related to heat or rain exposure, limited bathroom access, walking on some unpaved roads, roads with hills, curves, or construction work, as well as exposure to insects such as mosquitos, wildlife such as snakes, and flora or fauna such as poison oak or ivy. At any time, if you need a break, vehicles will be in nearby for easy access, extra hydration, and rest. There will also be vehicles to transport more significant injuries to appropriate medical resources. As a student, you can access the IHS health clinic services on campus free of charge.

<u>Alternative</u>: You will have the option to stay in the class, but you will not be asked to take the surveys.

<u>Benefits</u>: You may enjoy hearing traditional stories from elders and learning about drum making and other traditional activities, as well as enjoy gatherings where we share healthy foods. You might also like creating a digital story, film making, and going on field trips. You may learn new skills about leadership and how to have healthy relationships and behaviors. It might also make you feel proud to be a part of something that could help the health and wellness of Native American youth across the country.

<u>Compensation</u>: You will be paid up to \$75 in online gift cards for completing the online check-in surveys. You will receive \$20 for taking the second survey; \$25 for taking the third survey; and \$30 for taking the final survey.

#### Other Information

There are times when we may not be able to keep what we learn private. If you tell us that a child or elder is being abused, or if we think you are at risk of hurting yourself or someone else, we may need to report it. Also, sometimes government or university staff review studies to make sure they are being done safely and legally. If this study is reviewed, someone may look at the study records. The reviewers will protect your privacy. The study records will not be used to put you at risk of harm.

We will produce a report about the study. In the report we produce, we will not include any information that will make it possible to identify you or any other person. If you would like to see a copy of the final report once the study is finished, you can contact Dr. Tessa Evans-Campbell.

If you don't want to be in the study, you don't have to participate. Remember, being in this study is up to you and no one will be upset if you don't want to participate or even if you change your mind later and want to stop.

You can ask any questions about the study. If you have a question later, you can call me [insert your telephone number] or ask me next time.

Signing your name at the bottom means that you agree to be in this study. You have been given a copy of this form for you to keep.

| Researcher's signature | Date | |
|---|---|---|
| Your statement: | | |
| This research has been explained to me. I agree to questions. If I have more questions, I can ask the r | • | e to a |
| Your signature | <br>Date | |
| If you do not want to participate, please sign your | name below. | |
| If you do not want to participate, please sign your Your signature | name below. Date | |
| | <b>Date</b> f us about the study, please sign your name | |
| Your signature If you are unsure and would like to talk with one of | <b>Date</b> f us about the study, please sign your name | |